CLINICAL TRIAL: NCT03159091
Title: Multicenter Double-blind Placebo-controlled Parallel-group Randomized Clinical Trial of Efficacy and Safety of Rengalin in the Treatment of Cough in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Clinical Trial of Efficacy and Safety of Rengalin in the Treatment of Cough in Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Materia Medica Holding (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MMH-RN-005
Record Dates: First submitted 2017-05-17; First posted 2017-05-18 (Actual); Results first posted 2020-12-11 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2019-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rengalin (Experimental): Oral administration. Two tablets per intake. The tablet should be held in the mouth until complete dissolution. 2 tablets 3 times a day without food (i.e. 15-30 min prior to meal or 15-30 min after meal).
  Interventions: Drug: Rengalin
- Placebo (Placebo Comparator): Oral administration. Two tablets per intake. The tablet should be held in the mouth until complete dissolution. 2 tablets 3 times a day without food (i.e. 15-30 min prior to meal or 15-30 min after meal).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rengalin — Oral administration.
  Arms: Rengalin
Drug: Placebo — Oral administration.
  Arms: Placebo

SUMMARY:
The purpose of this study is to obtain additional data on efficacy and safety of Rengalin in the treatment of cough in patients with stable obstructive pulmonary disease

DETAILED DESCRIPTION:
Design: multicenter, double-blind, randomized, parallel group placebo-controlled study.

The study will enroll men and women (aged 40 to 80 years) with cough associated with stable chronic obstructive pulmonary disease (COPD). Subjects with COPD diagnosed more than 12 months earlier obtaining allowed basic therapy and retaining cough ≥2 points (according to cough severity scale [CSS]) despite their therapy should be considered as the study candidates.

After signing patient information leaflet (informed consent form) to participate in the clinical study, collection of medical history and objective examination are performed, cough severity is assessed (using CSS; at baseline evaluation of diurnal and nocturnal cough the number of episodes and cough severity in the preceding day is taken into account) as well as intensity of COPD effect on the subject (САТ test), concomitant therapy is recorded, computer spirometry with evaluation of baseline FEV1/FVC and post-bronchodilator FEV1 (where respiratory function cannot be assessed, the results of the previous examination dating no more than 3 months earlier may be used). Females of childbearing potential will undergo pregnancy test.

If a patient meets the inclusion criteria and does not demonstrate any of the exclusion criteria at Visit 1 (Day 1), he/she is randomized to one of 2 groups: group 1 patients will receive Rengalin at 2 tablets 3 times a day for 4 weeks; group 2 patients will receive placebo using Rengalin dosing regimen for 4 weeks.

The patient will be monitored for 4 weeks (screening, randomization - before day 1, treatment - 4 weeks). During follow-up period two visits are scheduled (Visit 1 (Day 1) and Visit 2 (Week 4) at which objective examination, recording cough severity (using CSS) will be carried out, COPD effect on the subjects (САТ test) and concomitant therapy will be evaluated. At Visit 2 (after 4-week treatment period) compliance will be additionally assessed.

At one of the clinical sites (Research Institute of Pulmonology, Russian FMBA), patients will be monitored for cough on a daily basis (using the WHolter™ monitor), with the data used as an additional measure to evaluate efficacy.

Subjects are allowed to take basic COPD therapy and medications for their co-morbidities in the course of the study, except for the medicines listed in "Prohibited concomitant treatment".

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both sexes aged from 40 to 80 years old.
2. COPD diagnosed (in accordance with the GOLD-2014 guidelines) ≥12 months before inclusion.
3. Stable course of COPD (≥ 6 weeks free of disease progression).
4. Mild, moderate or severe degree of bronchial obstruction (FEV1/FVC < 0.7; post-bronchodilator FEV1 ≥30% of predicted value).
5. CSS score ≥2.
6. Stable dose of standard therapy within the preceding 4 weeks.
7. Use of and adherence to contraceptive methods by fertile-age patients of both sexes during the study.
8. Availability of a signed patient information sheet (Informed Consent form) for participation in the trial.

Exclusion Criteria:

1. Earlier diagnosis of intra- or extrathoracic causes of cough (e.g., asthma, malignant neoplasm of lung, tuberculosis, sarcoidosis, α1-antitrypsin deficiency, bronchiectasis, cystic fibrosis, interstitial pulmonary diseases, perennial allergic rhinitis, gastro-oesophageal reflux disease, use of ACE inhibitors, disease of upper respiratory tract, etc.).
2. Cough associated with eating.
3. An exacerbation of COPD, acute upper and/or lower respiratory infection at inclusion or in the previous 4 weeks.
4. Modifications to standard drug therapy (dose escalation, replacement of medicines prescribed or addition of new medications) in the previous 4 weeks.
5. Very severe degree of bronchial obstruction (post-bronchodilator FEV1 <30% pred or < 50% and chronic respiratory failure).
6. Haemoptysis.
7. Stroke in the preceding 3 months or stroke with long-term residual neurological deficit within 6 months before study entry.
8. Acute coronary syndrome, myocardial infarction within 6 months before study enrollment.
9. Unstable or life-threatening arrhythmia in the previous 3 months.
10. Acute or chronic heart failure (NYHA (1964) Class III or IV).
11. Presence or suspicion of oncological disease.
12. Body Mass Index (BMI) ≤18 kg/m2 or ≥40 kg/m2.
13. Chronic kidney disease (categories С3-5 А3).
14. Hepatic failure (Child-Pugh class C)
15. Exacerbation or decompensation of a chronic disease that would affect the patient's ability to participate in the clinical trial.
16. For smokers - intention to quit smoking in the next 4 weeks.
17. Allergy/intolerance to any of the components of medications used in the treatment.
18. Course intake of medicines listed in the section 'Prohibited concomitant treatment' for 4 weeks prior to the enrollment in the trial.
19. Participation in other clinical trials within 3 months prior to the enrollment in this study.
20. Patients who, from investigator's point of view, will fail to comply with the observation requirements of the trial or with the dosing regimen of the investigational drug.
21. Other conditions preventing the patient from normal participation (e.g., planned business or other trips).
22. Drug addiction, alcohol use in the amount over 2 units of alcohol a day, mental diseases.
23. Pregnancy, breast-feeding, unwillingness to use contraception during the study.
24. Patient is related to the research staff of the clinical investigative site who are directly involved in the trial or is the immediate family member of the investigator. The immediate family members include husband/wife, parents, children or brothers (or sisters), regardless of whether they are natural or adopted.
25. Patient works for MATERIA MEDICA HOLDING company (i.e., is the company's employee, temporary contract worker or appointed official responsible for carrying out the research or their immediate family).

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2017-06-16 (Actual); Primary Completion 2019-04-25 (Actual); Study Completion 2019-04-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (18):
- Russia (18):
  - Regional state budgetary health care institution "Regional Clinical Hospital", Barnaul
  - Regional state budget health care institution "City Hospital No. 5, Barnaul", Barnaul
  - NUZ "Road Clinical Hospital at the station Chelyabinsk JSC" RZhD ", Chelyabinsk
  - The State Budget Health Institution "Regional Clinical Hospital No. 4", Chelyabinsk
  - Federal State Budgetary Educational Institution of Higher Education "Kazan Medical University"/Central City Clinical Hospital and Clinic #18, Kazan'
  - Federal State Budgetary Educational Institution of Higher Education "Kazan Medical University"/Professor's Clinic, Kazan'
  - Pirogov Russian National Research Medical University, Moscow
  - State Budgetary Institution of Health Care of the Nizhny Novgorod Region "City Clinical Hospital No. 10", Nizhny Novgorod
  - Ryazan State Medical University named after academician I.P. Pavlov, Ryazan
  - North-Western State Medical University named after I.I. Mechnikov, Saint Petersburg
  - North-western State Medical University named after I.I.Mechnikov, Saint Petersburg
  - St. Petersburg State Budgetary Public Health Institution "Vvedensky City Clinical Hospital", Saint Petersburg
  - The Federal State Institute of Public Health 'The Nikiforov Russian Center of Emergency and Radiation Medicine', Saint Petersburg
  - The First Pavlov State Medical University of St. Petersburg, Saint Petersburg
  - St. Petersburg State Budgetary Institution of Health "City Polyclinic No. 106", Saint Petersburg
  - Samara City Hospital №4, Samara
  - St. Petersburg State Budgetary Institution "City Hospital No. 40 in the Kurortny District", Sestroretsk
  - Voronezh Regional Clinical Hospital №1, Voronezh

REFERENCES:
- [Derived] Avdeev SN, Vizel AA, Abrosimov VN, Zaicev AA, Ignatova GL, Khamitov RF, Mikhaylusova MP, Shapovalova JS, Pavlysh EF, Trofimov BI, Emelyanov AV, Martynenko TI, Martynenko VA, Kostina NE, Chizhov DA, Chizhova OY, Kuzubova NA, Makova EV, Makarova EV. Management of Cough in Patients with Chronic Obstructive Pulmonary Disease: Results of the Multicenter Randomized Placebo-Controlled Clinical Trial. Int J Chron Obstruct Pulmon Dis. 2021 May 5;16:1243-1253. doi: 10.2147/COPD.S292109. eCollection 2021. PMID 33981141

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rengalin | Placebo
Started | 121 | 117
Completed | 116 | 113
Not Completed | 5 | 4
Not completed — Incorrect inclusion ineligible patient | 5 | 3
Not completed — Patient has taken no dose of study drug | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rengalin | Placebo | Total
Number analyzed (Participants) | 121 | 117 | 238
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (7.9) | 64.8 (8.4) | 64.3 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 23 | 50
  Male | 94 | 94 | 188
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Russia | 121 | 117 | 238

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With a Positive Treatment Response
Description: Cough Severity Scale (CSS) total score. Cough intensity according to the scale is assessed in daytime and at night in points where 0 - no cough, 5 - continuous exhausting cough in daytime and at night. Response criterion: ≥1 lower total CSS score compared to baseline.
Time Frame: in 4 weeks of the treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Rengalin | Placebo
Number analyzed (Participants) | 116 | 113
Participants | 97 | 82
Statistical Analysis 1: Comparison: Rengalin vs Placebo; Test type: Superiority; p = 0.0422, G-test (Chi-square)

2. Secondary Outcome: Severity of Cough After 4 Weeks Compared to Baseline
Description: Cough Severity Scale (CSS) total score. Cough intensity according to the scale is assessed in the daytime and at night in points, where 0 - no cough, 5 - continuous exhausting cough in the daytime, and at night.
Time Frame: Baseline and 4 weeks after the treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rengalin | Placebo
Number analyzed (Participants) | 116 | 113
score on a scale
  Initial total score | 4.18 (1.42) | 4.12 (1.42)
  Total score after 4 weeks | 2.56 (1.35) | 2.78 (1.16)
  ∆ between initial and 4 weeks total scores | 1.62 (1.38) | 1.35 (1.20)
Statistical Analysis 1: Comparison: Rengalin vs Placebo; This analysis applies to ∆ between initial and 4 weeks total scores row; Test type: Superiority; p = 0.1101, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Percentage of Patients With ≥50% Lesser Cough Severity at 4 Weeks
Description: Number of Participants with a Decrease from Baseline of ≥50% in Cough Severity at 4 weeks. Based on the total Cough Severity Scale (CSS) score. Cough intensity according to the scale is assessed in the daytime and at night in points, where 0 - no cough, 5 - continuous exhausting cough in the daytime and at night.
Time Frame: in 4 weeks of the treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Rengalin | Placebo
Number analyzed (Participants) | 116 | 113
Participants | 49 | 37
Statistical Analysis 1: Comparison: Rengalin vs Placebo; Test type: Superiority; p = 0.1373, G-test (Chi-square)

4. Secondary Outcome: Changes in Clinical Symptoms of Chronic Obstructive Pulmonary Disease (COPD)
Description: Based on the total COPD Assessment Test (CAT) score. CAT consists of 8 items. Each item ranges from "0" to "5" balls. The total score ranges from minimum "0" to maximum "40" points. Higher values represent a worse outcome.
Time Frame: in 4 weeks of the treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rengalin | Placebo
Number analyzed (Participants) | 116 | 113
score on a scale
  Initial total score | 19.9 (6.8) | 20.3 (6.6)
  Total score after 4 weeks | 16.6 (6.9) | 17.8 (6.8)
  ∆ between initial and 4 weeks total scores | 3.3 (4.2) | 2.5 (4.1)
Statistical Analysis 1: Comparison: Rengalin vs Placebo; Test type: Superiority; p = 0.0870, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Percentage of Patients With no Exacerbation of COPD
Description: COPD exacerbation is defined as an acute event characterized by aggravation of the event within 2-3 or more days. Exacerbation manifests in intensification of respiratory disorders beyond their regular daily fluctuations and require administration of products in addition to the previously prescribed basic therapy as well as a rescue drug for symptom relief (salbutamol). Additional products include antibacterial drugs, systemic corticosteroids and/or emergency therapy (ambulance call) or hospitalization for COPD exacerbation.
  COPD exacerbation is recorded as an adverse event. If a COPD exacerbation develops within the first week of the subject participation in the study, it will not be considered as a secondary inefficacy criterion
Time Frame: in 4 weeks of the treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Rengalin | Placebo
Number analyzed (Participants) | 116 | 113
Participants | 115 | 113
Statistical Analysis 1: Comparison: Rengalin vs Placebo; Test type: Superiority; p = 1.0, Fisher Exact

ADVERSE EVENTS:
Time Frame: 4 weeks (screening + randomization - up to 1 days, study therapy - 4 weeks).
Arm/Group | Rengalin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/121 | 1/116
Serious Adverse Events (participants affected / at risk) | 2/121 | 1/116
Other Adverse Events (participants affected / at risk) | 14/121 | 11/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rengalin (N=121) | Placebo (N=116)
Influenza A (H1N1) (Infections and infestations) | 1 (1) | 0 (0)
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rengalin (N=121) | Placebo (N=116)
Angular cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (1) — Stuck in the corners of the mouth.
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Labial herpes (Infections and infestations) | 0 (0) | 1 (1)
The rise in blood pressure (Vascular disorders) | 1 (1) | 0 (0)
Difficulty passing sputum (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Itchy palms (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Lumbar pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in the subscapularis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 2 (2)
Sleep disturbance (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) — Tinnitus on waking
Worsening hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
General weakness (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-17): https://cdn.clinicaltrials.gov/large-docs/91/NCT03159091/Prot_SAP_000.pdf